CLINICAL TRIAL: NCT02528565
Title: Laparoscopic Adjustable Gastric Banding With the Adhesix Bioring After Failed Gastric Bypass: a Prospective Evaluation in a High-volume Center
Brief Title: Gastric Banding After Failed Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-BA-01
Record Dates: First submitted 2015-07-15; First posted 2015-08-19 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with failed RYGB (EWL <50%)
  Interventions: Device: Adhesix Bioring

INTERVENTIONS:
Device: Adhesix Bioring

SUMMARY:
The safety and efficacy of the Adhesix Bioring adjustable gastric band will be assessed in patients after failed RYGB.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign the informed consent form prior to the index-procedure.
* Patient with failed RYGB defined as patients with EWL <50%.

Exclusion Criteria:

* Patient has a life expectancy of less than 2 year.
* Patient who is most likely expected not to be compliant with the proposed follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with failed RYGB receiving revisional LAGB.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage excess weight loss | 2 years

SECONDARY OUTCOMES:
Technical success defined as laparoscopic implantation of the Adhesix Bioring as intended by the surgeon without conversion to open repair. | During procedure
Complications (perioperative, early and late) | 2 years
Mortality | 2 years
Regression of co-morbidities | 2 years
BAROS score | 2 years
Frequency of revisions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dillemans, MD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- AZ Sint Jan Brugge, Bruges, Belgium